CLINICAL TRIAL: NCT05818319
Title: Cystic Fibrosis in the Kidney: Monitoring the Effectiveness of Elexacaftor/tezacaftor/ivacaftor in Urine After a Short Pause of Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CFPT29092022
Record Dates: First submitted 2023-03-28; First posted 2023-04-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis (CF); CFTR Gene Mutation
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: CF patients will perform a challenged urine bicarbonate test three times during this trial; 1) before, 2) during, and 3) after ETI therapy pause. Each test performance takes 90 min. and is accompanied by baseline blood sampling. First, a baseline urine sample is collected. Then the test person ingests 79 mg. NaHCO3/kg body weight dissolved in tap water (2,25 mL/kg body weight) together with the same amount of clean tap water. After 90 min. the test person delivers the second urine sample, and the test is completed. The test should preferably be performed between breakfast and lunch, at least one hour after intake of food. There should be at least three days between each test.
  CF patients will be randomly allocated to an ETI treatment pause for either 12, 36, or 60 hours. Treatment will be resumed immediately after the pause is finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 12 hours ETI pause (Other)
  Interventions: Other: 12 hours ETI pause
- 36 hours ETI pause (Other)
  Interventions: Other: 36 hours ETI pause
- 60 hours ETI pause (Other)
  Interventions: Other: 60 hours ETI pause

INTERVENTIONS:
Other: 12 hours ETI pause — Patients with CF are randomly allocated to ETI pause lasting 12 hours.
  Arms: 12 hours ETI pause
Other: 36 hours ETI pause — Patients with CF are randomly allocated to ETI pause lasting either 36 hours.
  Arms: 36 hours ETI pause
Other: 60 hours ETI pause — Patients with CF are randomly allocated to ETI pause lasting either 60 hours.
  Arms: 60 hours ETI pause

SUMMARY:
In cystic fibrosis (CF) renal base excretion is impaired, due to mutations in the Cystic Fibrosis Transmembrane Regulator (CFTR) gene, since CFTR function is crucial in regulation of the kidney's HCO3- excretion.

The investigators suggest that challenged urine HCO3- excretion is a biomarker of CFTR function, which can be used to evaluate the extent of CFTR dysfunction and the possible correcting effects of CFTR modulating therapy.

This study aims to evaluate changes in challenged urine HCO3- excretion in CF patients, who are currently in treatment with the triple CFTR modulator combination therapy, Elexacaftor/tezacaftor/ivacaftor (ETI), before, during, and after a short treatment pause.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age >17 years) CF patients.
* Normal kidney function estimated by eGFR>90.
* Adults capable of understanding and voluntarily consenting.

Exclusion Criteria:

* Critical acute illness.
* Severe lung disease (ppFEV1<40%).
* Adults not capable of understanding and voluntarily consenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference in cumulative urine bicarbonate excretion before, during, and after ETI pause. | At baseline, after 12/36/60 hours of therapy pause and after therapy is resumed.
  Challenged urine HCO3- test: Quantification of urine bicarbonate excretion after an acute oral NaHCO3 challenge before, under, and after ETI pause.
Link between changes in ETI plasma concentration and changes in urine bicarbonate excretion. | At baseline, after 12/36/60 hours of therapy pause and after therapy is resumed.
  Venous blood sampling: ETI plasma concentration measurement. Challenged urine HCO3- test: Quantification of urine bicarbonate excretion

SECONDARY OUTCOMES:
Link between plasma acid-base status and urine acid-base excretion. | At baseline, after 12/36/60 hours of therapy pause and after therapy is resumed.
  Venous blood sampling: Venous acid-base measurements.
Changes in plasma concentration of ETI during the trial. | At baseline, after 12/36/60 hours of therapy pause and after therapy is resumed.
  Venous blood sampling: ETI plasma concentration measurement.
Changes in acid-base and fluid status during the trial. | At baseline, after 12/36/60 hours of therapy pause and after therapy is resumed.
  Venous blood sampling: Venous acid-base and fluid measurements.
Changes in electrolytes during the trial. | At baseline, after 12/36/60 hours of therapy pause and after therapy is resumed.
  Venous blood sampling: Venous electrolyte measurements. Challenged HCO3- urine test: Urine electrolyte measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jens G. Leipziger, Principal Investigator — Department of Biomedicine, Aarhus University, Denmark; Majbritt Jeppesen, Principal Investigator — Department of Infectious Diseases, Aarhus University Hospital, Denmark
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Aarhus C, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berg P, Svendsen SL, Sorensen MV, Larsen CK, Andersen JF, Jensen-Fangel S, Jeppesen M, Schreiber R, Cabrita I, Kunzelmann K, Leipziger J. Impaired Renal HCO3- Excretion in Cystic Fibrosis. J Am Soc Nephrol. 2020 Aug;31(8):1711-1727. doi: 10.1681/ASN.2020010053. Epub 2020 Jul 23. PMID 32703846
- [Background] Berg P, Sorensen MV, Rousing AQ, Vebert Olesen H, Jensen-Fangel S, Jeppesen M, Leipziger J. Challenged Urine Bicarbonate Excretion as a Measure of Cystic Fibrosis Transmembrane Conductance Regulator Function in Cystic Fibrosis. Ann Intern Med. 2022 Nov;175(11):1543-1551. doi: 10.7326/M22-1741. Epub 2022 Nov 1. PMID 36315944